CLINICAL TRIAL: NCT02710539
Title: Randomized Comparison of Once-daily Fixed combiNation vErsus freE-drug cOmbination of Three aNtihypertensive Agents in arteriaL hYpertension (the ONE&ONLY Trial)
Brief Title: Once-daily Fixed Combination of Three Antihypertensive Drugs
Acronym: ONE&ONLY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 124/D/2016
Record Dates: First submitted 2016-03-04; First posted 2016-03-16 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Arterial Hypertension
Keywords: arterial hypertension; antihypertensive drugs
MeSH Terms: conditions — Hypertension | interventions — Perindopril; Indapamide; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Free combination (Active Comparator): Perindopril 10 mg/daily, indapamide 2,5 mg/daily, and amlodipine 10 mg/daily will be given according to a free combination strategy
  Interventions: Drug: perindopril, indapamide , amlodipine
- Tripliam (Active Comparator): fixed combination of perindopril 10 mg/daily, indapamide 2,5 mg/daily, amlodipine 10 mg/daily
  Interventions: Drug: Tripliam (perindopril, indapamide, amlodipine)

INTERVENTIONS:
Drug: perindopril, indapamide , amlodipine — Free combination of perindopril 10 mg, indapamide 2,5 mg, amlodipine 10 mg
  Other Names: Procaptan, Indapamide, Norvasc
  Arms: Free combination
Drug: Tripliam (perindopril, indapamide, amlodipine) — Fixed combination of perindopril 10 mg, indapamide 2,5 mg, amlodipine 10 mg
  Other Names: Fixed combination of Procaptan, Indapamide, Norvasc
  Arms: Tripliam

SUMMARY:
Randomized comparison of once-daily fixed combiNation versus free-drug combination of three antihypertensive agents in arterial hypertension

DETAILED DESCRIPTION:
The aim of this randomized study is to compare a once-daily fixed combination pill with a free-drug combination of three antihypertensive agents in arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

Patients with arterial hypertension resistant to monotherapy

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who reach target blood pressure | From baseline to the end of the 3-month study period
  How many patients have blood pressure within normal limits

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Gaudio, MD, Study Chair — Sapienza University
Locations (1):
- University La Sapienza, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marazzi G, Pelliccia F, Campolongo G, Cacciotti L, Massaro R, Poggi S, Tanzilli A, Di Iorio M, Volterrani M, Lainscak M, Rosano GM. Greater cardiovascular risk reduction with once-daily fixed combination of three antihypertensive agents and statin versus free-drug combination: The ALL-IN-ONE trial. Int J Cardiol. 2016 Nov 1;222:885-887. doi: 10.1016/j.ijcard.2016.07.163. Epub 2016 Jul 29. PMID 27522394